CLINICAL TRIAL: NCT02199028
Title: Evaluation of Glucose Sensor and Insulin Infusion Set Failures: Hyaluronidase Study
Brief Title: Hyaluronidase Effect on Infusion Set Life
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Bruce A. Buckingham, Principle Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 28949; JDRF 17-2013/471 (Other Grant/Funding Number: JDRF)
Record Dates: First submitted 2014-01-28; First posted 2014-07-24 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: hyaluronidase; infusion sets; insulin pump; Continuous glucose monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Hyaluronoglucosaminidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyaluronidase, Then Control (Experimental): Participants assigned to active treatment arm (Hylenex) for weeks 1 and 3.
  On weeks 1 and 3 (Hyaluronidase weeks) subjects injected 1 milliliter (ml) Hyaluronidase (150 units/ml) into the catheter hub prior to connecting the insulin infusion set on Day 1 and 3 of infusion set wear.
  On weeks 2 and 4 (control weeks) no Hyaluronidase was administered.
  Interventions: Drug: Hyaluronidase; Other: Control
- Control, Then Hyaluronidase (Experimental): Participants were first assigned to the control arm. They received active treatment (Hyaluronidase) on weeks 2 and 4.
  On weeks 1 and 3 (control weeks) no Hyaluronidase was administered.
  On weeks 2 and 4 (Hyaluronidase weeks) subjects injected 1 milliliter (ml) Hyluronidase (150 units/ml) into the catheter hub prior to connecting the insulin infusion set on Day 1 and 3 of infusion set wear.
  Interventions: Drug: Hyaluronidase; Other: Control

INTERVENTIONS:
Drug: Hyaluronidase — 150 units/ml - subjects injected 1 milliliter (ml) into the catheter hub prior to connecting the insulin infusion set on Day 1 and 3 of infusion set wear.
  Other Names: Hylenex
Other: Control — No hyaluronidase administered into insulin infusion set.

SUMMARY:
This research study examines the effect of hyaluronidase on the length of time of insulin infusion set wear. The aim of the study is to improve the length of time that an infusion set can be worn by infusing hyaluronidase directly into the insulin infusion site.

DETAILED DESCRIPTION:
The investigators would like to see if the use of hyaluronidase will improve insulin infusion set survival and improve the onset of insulin action. The investigators will also assess the accuracy of the Dexcom G4P sensors with extended site use beyond the 7 day FDA approved time frame.

The use of sensor information combined with the knowledge of infused insulin from pump therapy could potentially help us detect when an infusion set is beginning to fail. Information from the sensor function to the point of failure, and sensor function in response to Tylenol may allow us to develop special formulas to determine when a sensor is not working well. This will be very important for creating an artificial pancreas.

Thirty subjects will be enrolled. Fifteen patients from each of the two sites: Stanford University and University of Colorado.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes for at least one year and using an insulin pump for at least 3 months
2. Total daily insulin dose of at least 0.4 units/kg/day
3. The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.
4. Age 12 to 45 years
5. Hemoglobin A1c level less than or equal to 10%
6. Willingness to infuse 1 ml of hyaluronidase (Hylenex) into the insulin infusion set after insertion on day 1 and day 3 of the week they are assigned to use hyaluronidase
7. Willingness to use a Silhouette or Comfort insulin infusion set throughout the study. The set includes the Duo Infusion Tubing for infusion of hyaluronidase (Hylenex).
8. Willingness to eat the same breakfast each morning for the first two weeks of the study
9. Willing to take two 500mg tablets of Tylenol Regular Strength and monitor glucose levels at ½, 1, 2, 4, 6, and 8 hours later.
10. For females, not currently known to be pregnant
11. An understanding of and willingness to follow the protocol and sign the informed consent
12. Must be able to understand spoken or written English

Exclusion Criteria:

1. Diabetic ketoacidosis in the past 6 months
2. Severe hypoglycemia resulting in seizure or loss of consciousness in the 6 months prior to enrollment
3. Known tape allergies
4. Current treatment for a seizure disorder
5. Cystic fibrosis
6. Active infection
7. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:
8. Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's primary care giver (i.e., parent or guardian)
9. Presence of a known adrenal disorder
10. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
11. Abuse of alcohol
12. Use of an OmniPod insulin infusion pump
13. Pregnant or lactating females

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Buckingham, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel PJ, Benasi K, Ferrari G, Evans MG, Shanmugham S, Wilson DM, Buckingham BA. Randomized trial of infusion set function: steel versus teflon. Diabetes Technol Ther. 2014 Jan;16(1):15-9. doi: 10.1089/dia.2013.0119. Epub 2013 Oct 3. PMID 24090124
- [Background] Muchmore DB, Vaughn DE. Accelerating and improving the consistency of rapid-acting analog insulin absorption and action for both subcutaneous injection and continuous subcutaneous infusion using recombinant human hyaluronidase. J Diabetes Sci Technol. 2012 Jul 1;6(4):764-72. doi: 10.1177/193229681200600405. PMID 22920800
- [Background] Clausen TS, Kaastrup P, Stallknecht B. Effect of insulin catheter wear-time on subcutaneous adipose tissue blood flow and insulin absorption in humans. Diabetes Technol Ther. 2009 Sep;11(9):575-80. doi: 10.1089/dia.2009.0058. PMID 19764836
- [Derived] DeSalvo DJ, Ly TT, Wadwa RP, Messer L, Westfall E, Gopisetty D, Hanes S, von Eyben R, Maahs DM, Buckingham BA. Continuous Glucose Sensor Survival and Accuracy Over 14 Consecutive Days. Diabetes Care. 2016 Aug;39(8):e112-3. doi: 10.2337/dc16-0796. Epub 2016 May 23. No abstract available. PMID 27222506

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 30 subjects with Type 1 diabetes between 12-45 years were enrolled at 2 academic medical centers. 28 subjects completed the full 4 weeks of the study. 2 subjects discontinued for the study early. The last subject completed in March 2015.
Groups:
- Hylenex, Then Control: Participants assigned to active treatment arm (Hylenex) for weeks 1 and 3.
  On weeks 1 and 3 (Hylenex weeks) subjects injected 1 milliliter (ml) Hylenex (150 units/ml) into the catheter hub prior to connecting the insulin infusion set on Day 1 and 3 of infusion set wear.
  On weeks 2 and 4 (control weeks) no Hylenex was administered.
- Control, Then Hylenex: Participants were first assigned to the control arm. They received active treatment (Hylenex) on weeks 2 and 4.
  On weeks 1 and 3 (control weeks) no Hylenex was administered.
  On weeks 2 and 4 (Hylenex weeks) subjects injected 1 milliliter (ml) Hylenex (150 units/ml) into the catheter hub prior to connecting the insulin infusion set on Day 1 and 3 of infusion set wear.
Period: Week 1
Arm/Group | Hylenex, Then Control | Control, Then Hylenex
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Week 2
Arm/Group | Hylenex, Then Control | Control, Then Hylenex
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0
Period: Week 3
Arm/Group | Hylenex, Then Control | Control, Then Hylenex
Started | 14 | 15
Completed | 13 | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Week 4
Arm/Group | Hylenex, Then Control | Control, Then Hylenex
Started | 13 | 15
Completed | 13 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects between 12-45 years (inclusive) with clinical diagnosis of type 1 diabetes for at least one year, using an insulin pump for at least 3 months, and with an A1C less than 10%. 30 total subjects across two sites were enrolled and randomized the first week to either be in the control or experimental arm.
Groups:
- Hylenex, Then Control; Control, Then Hylenex: Participants were first assigned to the control arm. They received active treatment (Hylenex) on weeks 2 and 4.
  On weeks 1 and 3 (control weeks) no Hylenex was administered.
  On weeks 2 and 4 (Hylenex weeks) subjects injected 1 milliliter (ml) Hylenex (150 units/ml) into the catheter hub prior to connecting the insulin infusion set on Day 1 and 3 of infusion set wear.
- Total: Total of all reporting groups
Arm/Group | Hylenex, Then Control | Control, Then Hylenex | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.80552 (8.22924) | 30.06919 (8.33594) | 27.52718 (8.57883)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Duration of Insulin Infusion Set Wear as a Measure of the Effect of Hyaluronidase Treatment
Description: Average (mean) days of wear are presented for each group. A longer period of wear was considered a better outcome.
Time Frame: Up to 4 weeks
Population: Thirty subjects were enrolled in this study; 28 completed all scheduled visits. Therefore, 117 total weeks of infusion set wear were available for analysis including 58 hyaluronidase weeks and 59 standard weeks.
Measure: Mean (Standard Deviation); unit: Days of wear
Units Other Than Participants: week of infusion set wear
Groups:
- Hyaluronidase: Infuse 1mL Hyaluronidase at time of infusion set placement and again on Day 3
  Hyaluronidase: If assigned to hyaluronidase week, subjects will inject 1 milliliter (ml) Hylenex (150 units/ml) into the catheter hub prior to connecting the insulin infusion set. They will then give a catheter fixed prime of 0.7 cc to clear the infusion set of hyaluronidase. On the morning of day 3 during a Hyaluronidase week, a second dose of 1ml Hylenex (150 units/1ml) will be injected through the catheter hub prior to breakfast using the Duo Infusion Set Tubing. They will then reconnect their pump catheter and give a fixed prime of 0.7 cc to clear the infusion set of hyaluronidase.
- Control: Subjects will not receive Hyaluronidase during this week
Arm/Group | Hyaluronidase | Control
Number analyzed (Participants) | 30 | 30
Number analyzed (week of infusion set wear) | 58 | 59
Days of wear | 5.7 (1.7) | 5.4 (1.9)

2. Secondary Outcome: Maximum Glycemic Excursion
Description: The effects of hyaluronidase on post-prandial glucodymamic parameters is presented as the estimated glycemic excursion, a composite value which was calculated based on peak glucose concentration (Cmax), time to Cmax (Tmax), time to early half-maximal glucose concentration (t50%), time to late t50%, and area under the curve (AUC) of glucose concentrations at time intervals of 120 and 240 minutes, with or without hyaluronidase. Estimated glycemic excursion for a patient with Type 1 diabetes that is less than 80 mg/dL is considered acceptable.
Time Frame: Up to 24 hours post infusion
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Hyaluronidase | Control
Number analyzed (Participants) | 30 | 30
mg/dL
  Day 1 0-1 hour of infusion set | 43.5 (44.5) | 69.5 (47.4)
  Day 1 12-24 hours of infusion set | 36.9 (35.1) | 72 (48.8)
  Day 2 24-48 hours of infusion set | 56.4 (25.9) | 51.6 (32)

3. Secondary Outcome: Pain Tolerability of Hyaluronidase Injections
Description: Patients recorded pain experience at the infusion site (at time of injection and pain each day of wear) in subject diaries on a 0-5 pain scale (0 = no pain and 5 = worst pain imaginable).
  The number of diary entries are presented by scale category.
Time Frame: Up to 4 weeks
Population: Only participants in the Hyaluronidase injections group completed diary entries to track pain.
Measure: Number; unit: Diary entries
Units Other Than Participants: Diary Entries
Groups:
- Hyaluronidase Injections: Infuse 1mL Hyaluronidase at time of infusion set placement and again on Day 3
  Hyaluronidase: If assigned to hyaluronidase week, subjects will inject 1 milliliter (ml) Hylenex (150 units/ml) into the catheter hub prior to connecting the insulin infusion set. They will then give a catheter fixed prime of 0.7 cc to clear the infusion set of hyaluronidase. On the morning of day 3 during a Hyaluronidase week, a second dose of 1ml Hylenex (150 units/1ml) will be injected through the catheter hub prior to breakfast using the Duo Infusion Set Tubing. They will then reconnect their pump catheter and give a fixed prime of 0.7 cc to clear the infusion set of hyaluronidase.
Arm/Group | Hyaluronidase Injections
Number analyzed (Participants) | 30
Number analyzed (Diary Entries) | 107
Diary entries
  "0" on 0-5 pain scale | 58
  "1" on 0-5 pain scale | 34
  "2" on 0-5 pain scale | 11
  "3" on 0-5 pain scale | 4
  "4" on 0-5 pain scale | 0
  "5" on 0-5 pain scale | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during subject's participation in the study (screening to final visit). Adverse events were followed from onset to resolution.
Description: Adverse events were recorded during weeks of infusion set wear. In the study a total of 117 weeks of infusion set wear were available for analysis including 58 hyaluronidase weeks and 59 control weeks.
Groups:
- Hyaluronidase Week: Infuse 1mL Hyaluronidase at time of infusion set placement and again on Day 3
  Hyaluronidase: If assigned to hyaluronidase week, subjects will inject 1 milliliter (ml) Hylenex (150 units/ml) into the catheter hub prior to connecting the insulin infusion set. They will then give a catheter fixed prime of 0.7 cc to clear the infusion set of hyaluronidase. On the morning of day 3 during a Hyaluronidase week, a second dose of 1ml Hylenex (150 units/1ml) will be injected through the catheter hub prior to breakfast using the Duo Infusion Set Tubing. They will then reconnect their pump catheter and give a fixed prime of 0.7 cc to clear the infusion set of hyaluronidase.
- Control Week: Subjects will not receive Hyaluronidase during this week
Arm/Group | Hyaluronidase Week | Control Week
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 16/30 | 17/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyaluronidase Week (N=30) | Control Week (N=30)
Erythema >10 mm diameter (Skin and subcutaneous tissue disorders) | 16 (20) | 17 (19) — Erythema at infusion set insertion site
Infection at infusion set site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — abscess at insertion site
Infection at sensor site (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — abscess at Dexcom sensor insertion site
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Tape allergy from Dexcom sensor

LIMITATIONS AND CAVEATS:
This was a proof on concept pilot study and included a small number of participants. There was no evidence that hyaluronidase prolonged infusion set wear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No